CLINICAL TRIAL: NCT05760755
Title: Stick Together - a Dyadic Web-intervention for Younger Patients with Breast Cancer and Their Partners
Brief Title: Stick Together - Pilot Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Committee for Health Education (Other); TrygFonden, Denmark (Industry); Sygekassernes Helsefond (Other); Danish Cancer Society (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Annika von Heymann, Post.doc., Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P-2020-246; H-22032044 (Other: Videnskabsetisk Komité (RegionH))
Record Dates: First submitted 2023-01-26; First posted 2023-03-08 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Stick Together) (Experimental): Intervention group (all participants)
  Interventions: Behavioral: Stick Together

INTERVENTIONS:
Behavioral: Stick Together — The intervention consists of 12 online modules, completed flexibly during and immediately after primary cancer treatment. The intervention contains interviews with other couples, psychoeducational information, and interactive exercises on themes such as dyadic coping and communication, being diagnosed at a young age, fertility and children, and life after treatment.

SUMMARY:
This pilot study investigates the acceptability and feasibility of 'Stick Together', a self-guided online intervention, for younger women with breast cancer and their cohabiting partners.

DETAILED DESCRIPTION:
This one-arm feasibility study pilots the 'Stick Together' intervention among 20 women newly diagnosed with breast cancer at age 25-49 and their cohabiting partners. The intervention aims to strengthen couples' positive dyadic coping and communication, as well as participants mental health and quality of life, as well as quality of life of underage children.

ELIGIBILITY:
Inclusion Criteria (patients):

* women newly diagnosed with first primary breast cancer, treated with curative intent at Department of breast surgery, Gentofte Hospital
* living with a romantic partner

Inclusion Criteria (partners):

* living in romantic partnership with a patient eligible for the intervention

Exclusion Criteria (both patients and partners):

* severe relationship difficulties or current couples counselling
* severe, untreated mental illness in one or both partners
* capable of participating (mastery of Danish language, available smartphone, tablet or other device, no cognitive impairment)

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Participation (Acceptability 1) | baseline
  Percentage of eligible participants consenting to participate
Participants satisfaction (Acceptability 2) | Post-intervention follow-up (7-9 months post diagnosis)
  Percentage of participants satisfied with the intervention
Completion (Feasibility) | Post-intervention (7-9 months post diagnosis)
  Percentage of participants completing the intervention (65% completion)

SECONDARY OUTCOMES:
Change from baseline to post-intervention in supportive dyadic coping | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on supportive dyadic coping (min 5, max 25), as measured by the Dyadic coping inventory subscale. Higher scores indicate better outcome.
Change from baseline to post-intervention in delegated dyadic coping | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on delegated dyadic coping (min 2, max 10), as measured by the Dyadic coping inventory subscale. Higher scores indicate better outcome.
Change from baseline to post-intervention in negative dyadic coping | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on negative dyadic coping (min 4, max 20), as measured by the Dyadic coping inventory subscale. Higher scores indicate worse outcome.
Change from baseline to post-intervention in stress communication | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on stress communication (min 4, max 20), as measured by the Dyadic coping inventory subscale. Higher scores indicate better outcome.
Change from baseline to post-intervention in satisfaction with dyadic coping | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on satisfaction with dyadic coping (min 2, max 10), as measured by the Dyadic coping inventory subscale. Higher scores indicate better outcome.
Change from baseline to post-intervention in joint dyadic coping | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on joint dyadic coping (min 5, max 25), as measured by the Dyadic coping inventory subscale. Higher scores indicate better outcome.
Change from baseline to post-intervention in perceived stress | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on perceived stress (min 0, max 16), as measured by the Perceived Stress Scale. Higher scores indicate worse outcome.
Change from baseline to post-intervention in anxiety | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on anxiety symptoms (min 0, max 21), as measured by the Generalized anxiety scale-7. Higher scores indicate worse outcome.
Change from baseline to post-intervention in depression | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on depression symptoms (min 0, max 27), as measured by the Patient Health Questionnaire-9. Higher scores indicate worse outcome.
Change from baseline to post-intervention in protective buffering | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on protective buffering (min 8, max 40), as measured by the Ways of Giving Support-questionnaire subscale. Higher scores indicate worse outcome.
Change from baseline to post-intervention in active engagement | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on active engagement (min 5, max 25), as measured by the Ways of Giving Support-questionnaire subscale. Higher scores indicate better outcome.
Change from baseline to post-intervention in overprotection | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on overprotection (min 6, max 30), as measured by the Ways of Giving Support-questionnaire subscale. Higher scores indicate worse outcome.
Change from baseline to post-intervention in psychological quality of life | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on psychological quality of life (min 0, max 100), as measured by the World Health Organization Quality of Life Brief Version subscale (WHOQOL-BREF). Higher scores indicate better outcome.
Change from baseline to post-intervention in physical quality of life | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on physical quality of life (min 0, max 100), as measured by the World Health Organization Quality of Life Brief Version scubscale (WHOQOL-BREF). Higher scores indicate better outcome.
Change from baseline to post-intervention in social quality of life | Baseline, after intervention completion (average 8 months after diagnosis)
  Score on social quality of life (min 0, max 100), as measured by the World Health Organization Quality of Life Brief Version subscale (WHOQOL-BREF). Higher scores indicate better outcome.
Change from baseline to post-intervention in children's quality of life | Baseline, after intervention completion (average 8 months after diagnosis)
  Total mean score on quality of life (min 0, max 100), as measured by the Pediatric Quality of LIfe inventory (PEDSQL). Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of breast surgery, Gentofte Hospital, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared upon reasonable request to the Principal Investigator, when it can be allowed by applicable law and regulations.
Time Frame: Upon completion of study and publication of results.